CLINICAL TRIAL: NCT05930522
Title: Psychomotor Performance of Preterm Infants Born Between 24 and 35 Weeks of Gestation
Brief Title: Psychomotor Performance of Preterm Infants
Status: Completed | Type: Observational
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Other Study IDs: AWFiS/2023_3_PE
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-06

CONDITIONS: Psychomotor Development Impaired
Keywords: Preterm Birth; Preterm Infant; Motor abilities; Eurofit; Vienna test; Postural stability
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The first part involved 120 children in grades II and III of elementary schools. From this group, children were qualified for the second part of the study - 35 randomly selected children born on time (BoT) and 35 children born before 35 weeks of pregnancy (PB). EUROFIT tests, Vienna Tests and postural stability tests were carried out in both groups.

ELIGIBILITY:
Inclusion Criteria:

* preterm born (PB): born before 35 weeks of gestation
* both groups: aged 7-9 y during the research project

Exclusion Criteria:

* musculoskeletal injuries
* neurological disorders or other CNS damage

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 180 healthy school children
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Eurofit test | 20 minutes
  Motor abilities
Biodex Balance System SD | 15 minutes
  Static and dynamic postural stability
Vienna Test | 15 min minutes
  Speed reactions

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Ewertowska, PhD, Study Chair — Gdansk University of Physical Education and Sport
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided